CLINICAL TRIAL: NCT04346758
Title: Ultrasound-assisted Shamrock Method for Lumbar Plexus Nerve Block in Elderly Trauma Patients, Revisited.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Collaborators: University of Athens (Other)
Responsible Party: Principal Investigator, THEODOSIOS SARANTEAS, Associate Professor of Anesthesiology, Attikon Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AttikonH Shamrock 2019
Record Dates: First submitted 2019-11-21; First posted 2020-04-15 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Shamrock approach (Other): Patients undergoing orthopedic procedures of the lower extremeties are going to be studied. A modified Shamrock approach of the lumbar plexus is going to be used for postoperative analgesia, using an ultrasound-guided technique combined to a nerve stimulatior. The technique is going to be assessed as for accuracy, and safety.
  Interventions: Procedure: lumbar plexus block

INTERVENTIONS:
Procedure: lumbar plexus block — Patients undergoing orthopedic procedures of the lower extremeties are going to be studied. A modified Shamrock approach of the lumbar plexus is going to be used for postoperative analgesia, using an ultrasound-guided technique combined to a nerve stimulatior. The technique is going to be assessed as for accuracy, and safety.

SUMMARY:
A revised ultrasound-guided approach to the lumbar plexus is investigated as for efficacy and safety in elderly trauma patients undergoing operations of the lower extremeties.

DETAILED DESCRIPTION:
A modified ultrasound-guided Shamrock approach combined to nerve stimulation of the lumbar plexus is going to be investigated, in elderly trauma patients undergoing procedures of the lower extremities. The technique is going to be assessed as for its safety and its accuracy in localization of the plexus, by multiple measurements of the imaging time and needling time, In addition, efficacy and complications will be recorded and assessed during the immediate postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orthopedic trauma operations of the lower extremeties
* Age >70 years old

Exclusion Criteria:

* Preexisting neuropathy of Lumbar plexus
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up ie platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* Allergy to local anaesthetics
* Prior surgery at the lumbar region

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Time required to localize the lumbar plexus | 10 minutes (from the begining of imaging procedure) (time in seconds to localize the plexus)
  The time (in secondes) required of this modified Shamrock method to localize the lumbar plexus in the interpsoas compartment in elderly-trauma patients undergoing orthopedic procedures of the lower extremeties. Imaging time will be calculated (time to obtain appropriate imaging of the plexus) as well as needling time (time to obtain appropriate needle placement on the plexus)
Complications from lumbar plexus blockade | 1 month
  Safety of the modified Shamrock method of lumbar plexus blockade in elderly-trauma patients undergoing orthopedic procedures of the lower extremeties. All possible complications will be recorded (i.e. neurological complications, numbness, mobility disorder, haemmorhage, haematoma, e.t.c.)

SECONDARY OUTCOMES:
Postoperative pain | 4 hours (visual analogue scale 0-10 at 4 hours postoperatively)
  Postoperative pain relief 4 hours after completion of the block (visual analogue scale 0-10). A VAS score <4 is considered adequate.

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon Hospital, Athens, Greece